CLINICAL TRIAL: NCT00900211
Title: VORTEX-BIOBANK: Prospective Sample Collection for the VORTEX Randomised Radiotherapy Trial in Patients With Extremity Soft Tissue Sarcoma [VORTEX BIOBANK]
Brief Title: Tissue Sample Collection From Patients With Soft Tissue Sarcoma of the Arms, Hands, Legs, or Feet Treated on Clinial Trial CRUK-VORTEX
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Christie NHS Foundation Trust (Other)
Organization: National Cancer Institute (NCI) (NIH)
Other Study IDs: CDR0000581165; VORTEX-SA3002; VORTEX-REC-06/MRE03/3; ISRCTN76456502; EU-20795
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2013-08-26 (Estimated); Status verified 2008-04

CONDITIONS: Sarcoma
Keywords: recurrent adult soft tissue sarcoma; stage I adult soft tissue sarcoma; stage II adult soft tissue sarcoma; stage III adult soft tissue sarcoma; adult synovial sarcoma; adult angiosarcoma; adult epithelioid sarcoma; adult extraskeletal chondrosarcoma; adult leiomyosarcoma; adult liposarcoma; adult malignant fibrous histiocytoma; adult malignant hemangiopericytoma; adult malignant mesenchymoma; adult fibrosarcoma; adult neurofibrosarcoma
MeSH Terms: conditions — Sarcoma; Sarcoma, Synovial; Hemangiosarcoma; Chondrosarcoma, Extraskeletal Myxoid; Leiomyosarcoma; Liposarcoma; Histiocytoma, Malignant Fibrous; Hemangiopericytoma, Malignant; Malignant mesenchymal tumor; Fibrosarcoma; Neurofibrosarcoma | interventions — Microarray Analysis; Molecular Diagnostic Techniques

INTERVENTIONS:
Genetic: microarray analysis
Genetic: molecular diagnostic method
Other: biologic sample preservation procedure

SUMMARY:
RATIONALE: Collecting and storing samples of tumor tissue from patients with soft tissue sarcoma to test in the laboratory may help the study of cancer in the future.

PURPOSE: This laboratory is collecting tissue samples from patients with soft tissue sarcoma of the arms, hands, legs, or feet treated on clinical trial CRUK-VORTEX.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine early in the course of treatment which patients treated on clinical trial CRUK-VORTEX have an increased likelihood of distant metastases so as to highlight individuals who might benefit from early adjuvant systemic therapy.

OUTLINE: This is a multicenter study.

Tumour and normal tissue samples will be taken at the time of surgery during treatment on clinical trial CRUK-VORTEXand preserved for future microarray analyses. Tissue microarrays will be produced from both tumor and normal tissues. Blood samples will be collected for future DNA analysis.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed soft tissue sarcoma
* Receiving treatment on clinical trial CRUK-VORTEX
* Underwent surgery to remove the tumor no more than 3 months ago

PATIENT CHARACTERISTICS:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after completion of study treatment
* No other major medical illness that would preclude study treatment
* No other prior or concurrent malignancy except adequately treated nonmelanoma carcinoma of the skin or in situ carcinoma of the cervix

PRIOR CONCURRENT THERAPY:

* No prior radiotherapy to the local site
* No prior neoadjuvant or adjuvant chemotherapy

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2007-08; Primary Completion 2012-03 (Estimated)

PRIMARY OUTCOMES:
Increased likelihood of distant metastases

CONTACTS AND LOCATIONS:
Overall Officials: Catherine West, Study Chair — The Christie NHS Foundation Trust
Locations (12):
- United Kingdom (12):
  - Queen Elizabeth Hospital at University Hospital of Birmingham NHS Trust, Birmingham, England
  - Royal Orthopedic Hospital NHS Trust, Birmingham, England
  - Bristol Haematology and Oncology Centre, Bristol, England
  - Gloucestershire Oncology Centre at Cheltenham General Hospital, Cheltenham, England
  - Royal National Orthopaedic Hospital NHS Trust, Cheltenham, England
  - Middlesex Hospital, London, England
  - Christie Hospital, Manchester, England
  - Nottingham City Hospital, Nottingham, England
  - Cancer Research Centre at Weston Park Hospital, Sheffield, England
  - Robert Jones and Agnes Hunt Orthopaedic and District Hospital NHS Trust, Shropshire, England
  - Beatson West of Scotland Cancer Centre, Glasgow, Scotland
  - Glan Clwyd Hospital, Rhyl, Denbighshire, Wales